CLINICAL TRIAL: NCT01920191
Title: Phase I/II Study of Intradermal IMA950 Peptide-based Vaccine Adjuvanted With Intra Muscular Poly-ICLC in Combination With Temozolomide in Newly Diagnosed HLA-A2 Glioblastoma Patients
Brief Title: Phase I/II Trial of IMA950 Multi-peptide Vaccine Plus Poly-ICLC in Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: Immatics Biotechnologies GmbH (Industry); Oncovir, Inc. (Industry)
Responsible Party: Principal Investigator, Pierre-Yves Dietrich, Professor, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMA950 Poly ICLC
Record Dates: First submitted 2013-07-31; First posted 2013-08-09 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: CNS Tumor, Adult
Keywords: Glioblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma | interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMA 950 and Poly ICLC (Experimental)
  Interventions: Biological: IMA 950; Biological: Poly ICLC; Other: Immunomonitoring

INTERVENTIONS:
Biological: IMA 950
Biological: Poly ICLC
  Other Names: Hiltonol
Other: Immunomonitoring — Blood samples, DTH analysis

SUMMARY:
RATIONALE : IMA 950 is multi tumour-associated peptides (TUMAPs) vaccine, these peptides have been identified on primary glioblastoma multiforme (GBM) cells. Poly-ICLC is a potent vaccine adjuvant with broad innate and adaptive immune enhancing effects. IMA 950 and Poly-ICLC will be administered to patients alongside standard primary therapy for glioblastoma. This includes the alkylating drug temozolomide (TMZ). Effective vaccine-induced immune responses associated with prolonged survival have been observed in glioblastoma patients during TMZ adjuvant therapy, suggesting a possible synergistic effect. A second component of glioblastoma standard treatment is external beam irradiation of the tumor site post-surgery. As a side effect, potentially beneficial tumor-infiltrating immune cells may also be killed by radiation. However, the combination of radiation with immunotherapy has been suggested to be favorable both in pre-clinical models.

DETAILED DESCRIPTION:
OBJECTIVES

Primary

* Tolerability and safety of IMA950 adjuvanted with Poly-ICLC when given together with temozolomide, using CTCAE V 4.0.
* Immunogenicity of IMA950 plus Poly-ICLC when given together with temozolomide.

Secondary

* 6, 9 month progression free survival (PFS) using gadolinium enhanced MRI and clinical assessment according to revised RANO criteria
* Overall survival (OS)
* Immunologic endpoints (correlation between clinical and immunological responses):
* evaluation of peptide immunogenicity by tetramer staining
* analysis of memory, activation and homing marker expression by tetramer positive cells
* analysis of cytokine secretion and proliferation by antigen-specific CD4 and CD8 T cells
* analysis of the presence of T regulatory and myeloid-derived suppressor cells
* The immunological analyses will be performed on:
* peripheral blood mononuclear cells (PBMC)
* cultures of skin punch biopsy at delayed-type hypersensitivity (DTH) site
* tumor-infiltrating lymphocytes (TIL) if brain tissue is available at recurrence

OUTLINE

This is a monocentric, open label, one cohort, safety and immunogenicity, Phase I/II study.

A maximum of 16 HLA-A2 positive patients with newly diagnosed glioblastoma will be enrolled into the study after treatment with radiation therapy and concurrent temozolomide.

All patients will receive the same dose of IMA950 with Poly-ICLC and follow the same vaccination schedule which comprises a Vaccination Induction Phase of 4 intensive vaccinations, followed by a Vaccination Maintenance Phase of five vaccinations over a longer period.

The Vaccination Induction Phase will start a minimum of 7 days after the final radiotherapy/TMZ dose of CRT and 28 days (+7 days) prior to the first scheduled dose of adjuvant TMZ.

This will ensure that all 4 vaccinations in the Induction Phase will be administered a week after immunosuppressive therapy (i.e. combined radiotherapy and temozolomide) and will finish a week prior to the start of adjuvant TMZ.

Two Phases :

Induction phase, patient receive the first 4 doses of Poly ICLC mixed with IMA 950 Peptide based vaccine (subcutaneously or IM) on days 1,8,15, and 21 in absence of unacceptable toxicity or disease progression.

Maintenance Phase, patient receive Poly ICLC mixed with IMA 950 Peptide based vaccine (SC or IM) on day 21 of each adjuvant temozolomide cycle in absence unacceptable toxicity or disease progression.

Immunomonitoring assessments will be performed at 8 time points with blood samples collection and one DTH site analysis(after vaccination 5).

Brain MRI will be performed every two months for disease assessment.

N.B. :

An amendment has been accepted by Swissmedic and Local Ethics committee on september 2014, after suboptimal immunomonitoring preliminary assessments, the schedule of administration has been changed in order to improve the immunogenicity of the vaccine, as follows :

* injection of mixed peptides and adjuvant Poly ICLC
* 4 vaccinations in the induction phase instead of 6
* one site of injection (thigh)
* two arms for the next 10 patients to be included that will be equally divided in 2 groups : one group will be vaccinated subcutaneously and the other intramuscularly.

ELIGIBILITY:
Inclusion Criteria:

1. Histological documentation of glioblastoma. For experimental purposes only, 5 additional grade III astrocytoma may be included (these cases will not be included in the endpoints analysis).
2. Patients must have completed radiation therapy with concomitant temozolomide.
3. HLA-A2 positive.
4. Eastern Cooperative Oncology Group performance status of 0 or 1 (Appendix1).
5. Age > 18 years, life expectancy of least 4 months.
6. Patient must be on stable or decreasing dose of steroids, with a maximal dose of Dexamethasone of 4mg/day.
7. Adequate bone marrow, liver and kidney function.
8. Hepatitis B serology negative (HBcAg-seronegative)
9. Written (signed and dated) informed consent. Capable of co-operating with standard therapy and IMA950 with Poly-ICLC vaccinations and follow-up.

Exclusion Criteria:

1. Any other vaccination given within 2 weeks before first IMA950 vaccination.
2. History of cardiac disease: congestive heart failure > New York heart association class 2, active CAD, cardiac requiring anti-arrhythmic therapy or uncontrolled hypertension.
3. History of HIV infection or chronic hepatitis B or C or clinical active infections.
4. Patients with evidence of history bleeding diathesis.
5. Pregnant or potentially pregnant patients. Women of childbearing age must be tested for pregnancy (serum or urine HCG) before treatment and must not contemplate pregnancy during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Tolerability and safety of IMA950 adjuvanted with Poly-ICLC when given together with temozolomide, using CTCAE V 4.0 | up to 2 years

SECONDARY OUTCOMES:
6, 9 month progression free survival (PFS) using gadolinium enhanced MRI and clinical assessment according to revised RANO criteria | up to 2 years
Overall survival (OS) | up to 2 years
Immunologic endpoints | up to 2 years
  Correlation between clinical and immunological response. Blood sampling at baseline (week 4 and 5 after beginning of radiotherapy with concomitant temozolomide) and at week 10,11,12,16,19,23,27 and 31.
  Punch biopsy at DTH (Delayed Type Hypersensitivity) site performed 48h after DTH skin test 7 days after Vaccination 7.
  * evaluation of peptide immunogenicity by tetramer staining
  * analysis of memory, activation and homing marker expression by tetramer positive cells
  * analysis of cytokine secretion and proliferation by antigen-specific CD4 and CD8 T cells
  * analysis of the presence of T regulatory and myeloid-derived suppressor cells

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves Dietrich, Professor, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Centre of Oncology, Geneva, Switzerland

REFERENCES:
- [Derived] Migliorini D, Dutoit V, Allard M, Grandjean Hallez N, Marinari E, Widmer V, Philippin G, Corlazzoli F, Gustave R, Kreutzfeldt M, Blazek N, Wasem J, Hottinger A, Koka A, Momjian S, Lobrinus A, Merkler D, Vargas MI, Walker PR, Patrikidou A, Dietrich PY. Phase I/II trial testing safety and immunogenicity of the multipeptide IMA950/poly-ICLC vaccine in newly diagnosed adult malignant astrocytoma patients. Neuro Oncol. 2019 Jul 11;21(7):923-933. doi: 10.1093/neuonc/noz040. PMID 30753611